CLINICAL TRIAL: NCT02571946
Title: Feasibility of High Dose Proton Therapy in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis: Prospective Phase II Trial
Brief Title: Proton Beam Therapy in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Acronym: PTHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park Hee Chul, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-06-053
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Liver Neoplasm; Portal Vein Tumor Thrombosis; Proton Therapy
MeSH Terms: conditions — Liver Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Proton beam radiotherapy
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton beam therapy (Experimental)
  Interventions: Radiation: Proton beam therapy

INTERVENTIONS:
Radiation: Proton beam therapy

SUMMARY:
The standard treatment of advanced hepatocellular carcinoma (HCC) is sorafenib. Though the agent showed clear survival benefit in two randomized phase III trials, the benefit was modest and response rate was just a few percent. Therefore, other loco-regional modalities, like trans-arterial chemo-embolization (TACE), hepatic arterial infusion chemotherapy (HAIC), and radiotherapy (RT) were continuously tried, especially in locally advanced HCC including portal vein tumor thrombosis (PVTT).

With the advancement of conformal RT techniques, RT was actively applied in HCC, especially in PVTT combined HCC. Many researchers reported that there is a relationship between RT dose and tumor response rate. RT dose, however, is frequently limited because the complications (like radiation induced liver disease (RILD), radiation induced gastro-duodenal toxicity, etc.) are also closely related with higher exposed RT dose.

Proton beam has characteristic depth-dose distribution contrast to photon, the "Bragg peak". The advantage of this dose distribution could be more highlighted in HCC management, because of the weakness and maintenance importance of liver function itself in HCC patients. In fact, the superior results of proton beam therapy in HCC were constantly reported in several groups as prospectively as well as retrospectively.

In those background, the investigators planned the present study to evaluate the efficacy and safety of proton beam therapy in HCC patients combined with PVTT.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma (HCC) patients
* pathologically proven
* HCC diagnosed based on American Association for the Study of Liver Diseases (AASLD) guideline
* Portal vein tumor thrombosis (main, first branch, segmental)
* Discussion in tumor board including gastroenterologist, radiologist, radiation oncologist
* 20 or more age
* Eastern Cooperative Oncology Group performance status 0 to 2 within 1 week before participate
* Adequate bone marrow function (absolute neutrophil count ≥ 1.0 x 109/l, platelet ≥ 30 x 109/l, hemoglobin ≥ 8 g/dl)
* Adequate liver/renal function within 1 week before participate
* Child-Pugh class A, B, or early C (score ≤ 10)
* Total bilirubin <3.0 mg/dL, Prothrombin time/International normalized ratio <1.7, Albumin≥2.8g/dL, Aspartate aminotransferase/alanine aminotransferase<6 times of upper normal limit
* Serum creatinine < 1,5 x upper normal limit, glomerular filtration rate > 50 ml/min Informed consent
* Women of childbearing potential and male participants must agree to practice adequate contraception while on study and for at least 6 months following the last dose of RT and for at least 28 days following the last dose of sorafenib (whichever is later).

Exclusion Criteria:

* Uncontrolled hepatic encephalopathy
* Previous history of upper abdominal radiotherapy
* Status of pregnancy or breast feeding
* Less than 12 weeks of expected survival
* Uncontrolled ascites
* Combined with disease known as radiosensitive disorder (connective tissue disorder, Ataxia-telangiectasia)
* Hard to maintain stable respiration less than 5 minutes related with respiratory disease
* Combined with uncontrolled severe acute disease other than liver

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
one-year overall survival | one-year after proton beam therapy

SECONDARY OUTCOMES:
1 month objective response rate | 1 month after proton beam therapy
3 month objective response rate | 3 months after proton beam therapy
1 month portal vein tumor thrombosis response rate | 1 month after proton beam therapy
3 month portal vein tumor thrombosis response rate | 3 month after proton beam therapy
1 year progression free survival | one-year after proton beam therapy
1 year local progression free survival | one-year after proton beam therapy
1 year portal vein tumor thrombosis progression free survival | one-year after proton beam therapy
Adverse event | one-year after proton beam therapy
1 month Quality of life assessment compared with baseline | 1 month after proton beam therapy
3 month Quality of life assessment compared with baseline | 3 month after proton beam therapy
6 month Quality of life assessment compared with baseline | 6 month after proton beam therapy
Indocyanine green test change compared with baseline | 3 month after proton beam therapy
Hepatobiliary phase signal change after proton beam therapy | 3 month after proton beam therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea